CLINICAL TRIAL: NCT06444113
Title: A Phase IV, Prospective, Multicenter, Open-label, Mother-milk Study to Evaluate Ofatumumab Concentration in the Breast Milk of Lactating Women With Relapsing Forms of Multiple Sclerosis Receiving Ofatumumab
Brief Title: Concentration of Ofatumumab in the Breast Milk of Lactating Women With Relapsing Forms of Multiple Sclerosis
Acronym: KATHAROS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COMB157G2410; 2023-505283-11-00 (Other: CTIS)
Record Dates: First submitted 2024-05-30; First posted 2024-06-05 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
Keywords: Lactating women,; multiple sclerosis (MS); ofatumumab; milk concentration; breastfed infant
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ofatunumab (Experimental): Recommended dose as per ofatumumab label. Injection at weeks 0,1,2 and monthly starting at week 4.
  Interventions: Drug: Ofatunumab

INTERVENTIONS:
Drug: Ofatunumab — No study-treatment is provided for this study. Study participants will be treated with commercially available ofatumumab according to the local label.

SUMMARY:
This study will evaluate whether ofatumumab is excreted at quantifiable levels and at which concentrations in breast milk of lactating women with RMS). The study will include lactating mothers who plan to breastfeed and initiate/re-initiate ofatumumab 2-24 weeks post-partum.

DETAILED DESCRIPTION:
This is a Phase IV study in which breastfeeding mothers treated with ofatumumab and their babies are taking part for up to 1 year. The study consists of a Core Part and a Safety Follow-up Part. The Core Part includes a Screening period and a Sampling period. During the Screening period (up to 4 weeks), the study doctor will assess if mothers can join the study. The Sampling period, during which milk samples and a blood sample will be collected, will last for up to 12 weeks. The Safety Follow-up Part will last for about 9 months, to follow up on health and safety of mothers and their babies.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent must be obtained before any study assessment is performed.
2. Participant is female with a relapsing form of MS and at least 18 years of age at the time of providing consent.
3. Participant must be postpartum at the time of enrollment, plan to be exclusively breastfeeding and willing to provide breast milk samples.
4. Participant has delivered term infant (at least 37 weeks gestation).
5. Participant must plan to initiate or re-initiate or have initiated or re-initiated treatment with ofatumumab between 2 to 24 weeks postpartum. The decision to be treated with ofatumumab and to breastfeed is made in accordance with the treating physician and must be completely independent of the decision to participate in this study.

Exclusion Criteria:

1. Use of any investigational drugs within 5 half-lives of enrollment, or within 30 days or until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
2. Participant taking medications prohibited by the study protocol at screening.
3. Pregnant woman, confirmed by positive serum pregnancy test during screening.
4. Female of childbearing potential should use effective contraception as per local label.
5. Participant has history of chronic alcohol abuse or drug abuse in the last year.
6. Participant has any medical, obstetrical, psychiatric or other medical condition that, in the opinion of the Investigator, can jeopardize or would compromise the subject's ability to participate in this study or confound the study assessment.
7. Participant has history of breast implants, breast augmentation, or breast reduction surgery.
8. Participant has received anti-CD20 agents during the second and third trimesters of pregnancy.
9. Active infections, including mastitis (participant may be included once the infection is resolved).
10. Prior or current history of primary or secondary immunodeficiency, or participant in an otherwise severely immunocompromised state.
11. Participant with active hepatitis B disease prior to the initiation or re-initiation of ofatumumab. (Participant with positive hepatitis B serology should consult a liver disease medical standards to prevent hepatitis B reactivation.)
12. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
13. Any contraindication as per local label.
14. Participant who has an infant with any abnormality that may interfere with breastfeeding or confound the study assessment in the opinion of the Investigator.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-11-25 (Actual); Primary Completion 2026-05-18 (Estimated); Study Completion 2027-02-23 (Estimated)

PRIMARY OUTCOMES:
Concentration of ofatumumab in breast milk. | (pre-dose) on the day of second (or subsequent) maintenance dose, then 7, 14, 21, 28 days after the second (or subsequent) maintenance dose"
  Quantification of ofatumumab concentration in breast milk of lactating women with RMS who have initiated or re-initiated ofatumumab treatment post-partum.

SECONDARY OUTCOMES:
Evaluate other PK parameters of ofatumumab in breast milk and plasma of lactating women with RMS who have initiated or re-initiated ofatumumab treatment post-partum | 28 days after second(or subsequent) maintenance dose.
  proportion of at least one sample with quantifiable concentration; Maximum concentration; exposure (Area under curve); milk/plasma ratio
Estimation of relative infant dose of ofatumumab | 28 days after second (or subsequent) maintenance dose.
  Estimated relative infant dose (RID, %) over 28 days after the lactating mother receives second or subsequent maintenance dose
Safety data collected in lactating women receiving ofatumumab and their breastfed infants | Upto 12 months
  Rate and nature of adverse events in the mothers treated with ofatumumab to up to 12 months after ofatumumab treatment initiation/re-initiation Rate and nature of serious adverse events and any infection adverse events in the breastfed infants of mothers up to 12 months after ofatumumab treatment initiation/re-initiation
Plasma Pharmacokinetics of OMB157(Cmax) | over 28 days after the second (or any subsequent) maintenance dose.
  Maximum concentration (Cmax) of ofatumumab in breast milk over 28 days after the second (or any subsequent) maintenance dose.
Plasma Pharmacokinetics of OMB157(AUC) | over 28 days
  The exposure (area under the curve (AUC) of ofatumumab in milk over 28 days (from the second or any subsequent maintenance dose to the next maintenance dose after initiation or re-initiation of ofatumumab post-partum)
Plasma Pharmacokinetics of OMB157 (M/P Ratio) | at 28 days after the second or any subsequent maintenance dose.
  Milk/Plasma (M/P) ratio of ofatumumab at 28 days after the second or any subsequent maintenance dose.

CONTACTS AND LOCATIONS:
Locations (22):
- United States (5):
  - UCSF, San Francisco, California
  - UC Health Neuroscience Ctr, Aurora, Colorado
  - Northwestern Medicine Northwestern University, Winfield, Illinois
  - Brigham and Womens Hospital, Brookline, Massachusetts
  - Duke Neurology, Durham, North Carolina
- Germany (4):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Bochum
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Tübingen
- Italy (3):
  - Novartis Investigative Site, Foggia, FG
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Kielce
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Rzeszów
  - Novartis Investigative Site, Zabrze
- Caribbean Center for Clinical Research, Inc, Guaynabo, Puerto Rico
- United Kingdom (4):
  - Novartis Investigative Site, Cambridge
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Oxford
  - Novartis Investigative Site, Salford

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com.